CLINICAL TRIAL: NCT00969072
Title: A Long-term Extension Study of GI198745 in Subjects With Benign Prostatic Hyperplasia
Brief Title: Extension Study of GI198745 to Treat Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARI30016
Record Dates: First submitted 2009-07-23; First posted 2009-08-31 (Estimated); Last update posted 2010-09-13 (Estimated); Status verified 2010-09

CONDITIONS: Benign Prostatic Hyperplasia; Prostatic Hyperplasia
Keywords: GI198745; Long term extension study; BPH
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- GI198745 (Experimental)
  Interventions: Drug: GI198745 0.05mg; Drug: GI198745 0.5mg; Drug: GI198745 2.5mg

INTERVENTIONS:
Drug: GI198745 0.05mg — GI198745 (drug) - benign prostatic hyperplasia
Drug: GI198745 0.5mg — GI198745 (drug) - benign prostatic hyperplasia
Drug: GI198745 2.5mg — GI198745 (drug) - benign prostatic hyperplasia

SUMMARY:
The primary objective is to assess the safety of GI198745 0.05mg, 0.5mg, 2.5mg once daily for 52 weeks.

DETAILED DESCRIPTION:
Upon completion of 24 weeks of GI198745 0.05 mg, 0.5 mg, 2.5 mg, or placebo therapy in study ARI20005, subjects are enrolled into an extension phase and are continued on the same therapy once daily for up to further 28 weeks, followed by up to 16 weeks of post-dosing assessments.

ELIGIBILITY:
Inclusion Criteria:

* Has been receiving the investigational product for at least 20 weeks in the preceding dose finding study and the investigator or subinvestigator has confirmed the tolerability and has judged as appropriate to participate continuously in further 28 weeks treatment.

Exclusion Criteria:

* Is withdrawn from the dose finding study.
* Has less than 75% compliance with the investigational product in the dose finding study at given the informed consent for the long-term extension study.
* Has a prostate cancer at giving informed consent for participating in the long-term extension study; or is suspected to have a prostate cancer in palpation, ultrasound imaging, biopsy, etc. at giving informed consent for participating in the long-term extension study.
* Has the post void residual volume > 250 ml at starting the long-term extension study. (as measured by suprapubic ultrasound).
* Has chronic bacterial prostatitis or chronic urinary tract infections during the dose finding study
* Has acute urinary retention in the dose finding study.
* Has a history or current evidence of drug or alcohol abuse during the dose finding study
* Has been treated with any investigational product including post-marketing clinical trials during the dose finding study.
* Has myocardial infarction, coronary arterial bypass surgery, unstable angina, arrhythmia, congestive heart failure, cerebrovascular accident during the dose finding study.
* Has any concurrent disease or complication that, in the opinion of the investigator/sub-investigator, is difficult to evaluate efficacy of GI198745 in this study and that might poses additional risk to the patient.
* Is actively trying to procreate in the study period.
* Is unsuitable for this study, in the opinion of the investigator/sub-investigator.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2003-08; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
adverse events, laboratory test values (hematology, serum chemistry, electrolyte, and urinalysis), prostate specific antigen (PSA), vital signs (blood pressure, pulse rate), and post-void residual volume. | a 28-week extension treatment in the subjects entered into the 24-week dose finding study (ARI20005: multicentre, double-blind, randomised, placebo-controlled, parallel-group)

SECONDARY OUTCOMES:
prostate volume, symptom scores (IPSS), maximum urinary flow (Qmax), serum dihydrotestosterone (DHT), and testosterone | a 28-week extension treatment in the subjects entered into the 24-week dose finding study (ARI20005: multicentre, double-blind, randomised, placebo-controlled, parallel-group)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline